CLINICAL TRIAL: NCT02988336
Title: Thyromental Height Test as a New Method for Prediction of Difficult Intubation With Double Lumen Tube
Brief Title: TMHT - New Method of Difficult Intubation Prediction
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: TMHT-01
Record Dates: First submitted 2016-11-30; First posted 2016-12-09 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Airway Management; Predictive Value of Tests
Keywords: difficult intubation; thyromental height

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the usefulness of the Thyromental Height Test in prediction of difficult intubation using double lumen endotracheal tubes in patients scheduled for elective thoracic procedures.

DETAILED DESCRIPTION:
Proper prediction of the occurrence of difficult intubation plays a crucial role in anaesthesiology. For years attempts have been made to develop methods allowing anaesthesiologists to correctly predict the occurrence of difficult intubation. None of the currently used tests and anthropometric measurements present satisfying predictive value. Recent studies show promise in Thyromental Height Test (TMHT), which base on the height between the anterior borders of the mentum and the thyroid cartilage, measured while the patient lies in the supine position with closed mouth, as a single, non-invasive predictor of difficult intubation. Use of double lumen endotracheal tubes during thoracic procedures, due to greater diameter of the tube, may lead to higher occurrence of difficult intubation. That is why, the purpose of this study is to assess the usefulness of the TMHT in prediction of difficult intubation using double lumen endotracheal tubes in patients scheduled for elective thoracic procedures and relate it to other, commonly used predictive tests.

During routine, preoperative anaesthetic visit thyromental height, thyromental distance, sternomental distance and Mallampati scale score are assessed. Then, during direct laryngoscopy and intubation, score in Cormack-Lehane scale and occurrence of difficult intubation are noted.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective thoracic procedures, requiring general anaesthesia, direct laryngoscopy and intubation with a Robertshaw type double lumen endotracheal tubes
* consent for participation in the trail
* older than 18

Exclusion Criteria:

* emergency procedures
* visible anatomic abnormalities
* patients scheduled for awake fibre optic intubation
* lack of consent for participation in the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing elective thoracic procedures in university hospital, requiring general anaesthesia, elective direct laryngoscopy and intubation with a double lumen endotracheal tubes.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Thyromental height | immediate
  The height between the anterior border of the thyroid cartilage (on the thyroid notch just between the 2 thyroid laminae) and the anterior border of the mentum (on the mental protuberance of the mandible), in supine position with mouth closed, measured with a depth gauge, measured during routine preoperative anaesthetic visit.

SECONDARY OUTCOMES:
Thyromental distance | immediate
  The distance between the thyroid prominence and the most anterior part of the mental prominence of the mandible, measured with a standard centigrade ruler as the distance in centimetres with the patient in supine position, head fully extended, mouth closed, during routine preoperative anaesthetic visit.
Sternomental distance | immediate
  The distance in centimetres between the superior border of the manubrium sterni and the bony point of the mentum, with the patient in supine position, head fully extended, mouth closed, measured with a standard centigrade ruler, during routine preoperative anaesthetic visit.
score in modified Mallampati test | immediate
  The oropharyngeal view is assessed in sitting position, mouth maximally opened, tongue protruded, without phonation, measured during routine preoperative anaesthetic visit.
score in Cormack-Lehane scale | immediate
  During direct laryngoscopy the patient is graded in Cormack-Lehane Scale by the laryngoscopist.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiołek, MD PhD, Study Chair — School of Medicine with the Division of Dentistry in Zabrze. Medical University of Silesia. Department of Anaesthesiology and Critical Care.
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palczynski P, Bialka S, Misiolek H, Copik M, Smelik A, Szarpak L, Ruetzler K. Thyromental height test as a new method for prediction of difficult intubation with double lumen tube. PLoS One. 2018 Sep 13;13(9):e0201944. doi: 10.1371/journal.pone.0201944. eCollection 2018. PMID 30212462